## **DEPARTMENT OF PSYCHIATRY**

NEUROSCIENCES BUILDING WARNEFORD HOSPITAL OXFORD OX3 7JX, U.K. www.psych.ox.ac.uk

<u>Principal Investigator</u>: Prof Catherine Harmer <u>Email</u>: catherine.harmer@psych.ox.ac.uk

Tel: +44 (0)1865 618326

**<u>Primary Researcher</u>**: Michael Colwell, DPhil Student

Tel: +44 (0)1865 618 303

Email: michael.colwell@psych.ox.ac.uk





Participant Consent Form – The effect of seven day fenfluramine administration on cognition in healthy volunteers

**Document originally created:** 19/11/2020; Last update: 28/07/2021

## **PARTICIPANT CONSENT FORM**

CUREC Approval Reference: R69642/RE001

## The effect of seven day fenfluramine administration on cognition in healthy volunteers

Purpose of Study: To investigate the effects of fenfluramine on cognitive ability, comparing the effects of the drug with placebo.

| | | Please initial each<br>box |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet version dated for the above study. I have had the opportunity to consider the information carefully, ask questions and have had these questions answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without any adverse consequences or academic penalty. | |
| 3 | I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. | |
| 4 | I have been advised as to what I need to do for this research (especially with regard to drug intake) and I agree to follow the instructions given to me. | |
| 5 | I understand that blood and urine samples will be taken to assess my eligibility criteria for the study. I understand my urine sample will used to assess pregnancy status (if appropriate) and current drug use. I understand my blood samples will be used as standard screening to check physical health (liver function, urea, and electrolytes. I understand that the samples will be destroyed after completion of the eligibility assessment, or if I withdraw my consent. | |
| 6 | I understand that saliva samples will be taken during the study and that these samples will be tested for cortisol levels. I understand that the samples will be destroyed after study has ended, or if I withdraw my consent. | |
| 7 | To the best of my knowledge, I do not meet any of the exclusion criteria outlined in the information sheet for this research. If this changes at a later date during study participation, I agree to notify the researchers immediately. | |

| 8 | | ~ | dy may be looked at by designated permission for these individuals to |
|---|---|---|---|
| 9 | I understand who will have stored and what will happ | · | data provided, how the data will be end of the project. |
| 10 | I consent to answering sc part. | reening questions to o | confirm my eligibility to take |
| 11 | including those working o | outside of the UK and | ared with other researchers,<br>the EU, to be used in other research<br>be anonymised so that I cannot be |
| 12 | I understand how this res | earch will be written | up and published. |
| 13 | I understand that this project has been reviewed by, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. | | |
| 14 | I understand how to raise | a concern or make a | complaint. |
| 15 | | understand that all information will be kept strictly confidential except in the are circumstance in which it is judged that I, or someone else, is at immediate isk of serious harm. | |
| 16 | I understand that I have been advised not to drink alcohol or carry out activities requiring full alertness (such as driving) during the week of drug/placebo administration if I am aware of any impairment. | | |
| 17 | I agree to take part in the study | | |
| Optional: | contacting me about futu | ntact details to be kept in a secure database for the purpose of bout future studies. I understand that agreeing to be contacted ne to participate in any further studies. | |
| Name of F | Participant | dd / mm / yyyy<br>Date | <u>Signature</u> |
| Name of p | person taking consent | dd / mm / yyyy<br>Date | <u></u> |